CLINICAL TRIAL: NCT03405558
Title: Effects of an Individually Tailored Endurance Training on the Performance Developement of Patients With Paraplegia During First Rehabilitation: an Observational Study
Brief Title: Performance Developement of Patients With Paraplegia During First Rehabilitation
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2017-01
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — As this is an observational study, we will only supervise testing and training sessions which were performed anyway during first rehabilitation as daily therapeutic routine

SUMMARY:
A high physical fitness is crucial for a good quality of life in persons suffering from a spinal cord injury. The aim of the present observational study is to investigate the influence of an individually tailored 8-week endurance training program on endurance performance of patients with a paraplegia during their first rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* male or female, paraplegia (AIS A-C, lesion Level Th1-Th12)
* Age 18-65 years
* Manual wheelchair user
* Patient during first rehabilitation

Exclusion Criteria:

* BMI ≥ 30
* unable to use an arm-crank Ergometer due to e.g. spasticity
* physical impairment, which makes it impossible to perform an arm-crank ergometry
* Progressive disease (g.g. tumor, MS)
* Ventilator dependent
* existing cardiopulmonary disease
* Unstable medical situation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a paraplegia during the first rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Peak power | 10min
  Maximal performance reached during incremental exercise on an arm-crank ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No